CLINICAL TRIAL: NCT02329678
Title: Efficacy of Guided Tissue Regeneration Membrane in the Healing of Apicomarginal Defects - A Prospective, Controlled Clinical Trial.
Brief Title: Efficacy of Guided Tissue Regeneration Membrane in the Healing of Apicomarginal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Professor, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pgimsrohtak
Record Dates: First submitted 2014-12-17; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Apicomarginal Defects
Keywords: Apicomarginal defects; clinical study/trial; collagen membrane; guided tissue regeneration; endodontic microsurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- collagen membrane group and control group (Active Comparator): GTR group: a bioresorbable collagen membrane (Healiguide, Advanced Biotech Products (P) Ltd., Encoll Corp., Fremont, CA, USA) was placed over the apicomarginal defect, covering 2-3mm of the healthy bone around all the margins after periodical surgery.
  Interventions: Procedure: Peripical surgery
- Control group (Active Comparator): Control Group:No membrane was placed after periapical surgery.
  Interventions: Procedure: Peripical surgery

INTERVENTIONS:
Procedure: Peripical surgery — Thirty patients meeting inclusion criteria were selected and allocated randomly into two groups: collagen membrane group and control group. Clinical and radiographic measurements were recorded during follow up at regular intervals of 0, 3, 6, 9, and 12 months after surgery. The criteria for success included the absence of clinical signs and symptoms, and complete or incomplete radiographic healing.

SUMMARY:
Introduction: The present clinical trial was conducted to evaluate the efficacy of membrane barrier in the healing of apicomarginal defects.

Methods: Thirty patients meeting inclusion criteria were selected and allocated randomly into two groups: collagen membrane group and control group. Clinical and radiographic measurements were recorded during follow up at regular intervals of 0, 3, 6, 9, and 12 months after surgery. The criteria for success included the absence of clinical signs and symptoms, and complete or incomplete radiographic healing.

DETAILED DESCRIPTION:
Title: Efficacy of guided tissue regeneration membrane in the healing of apicomarginal defects - A prospective, controlled clinical trial.

Apicomarginal defects, localized bony defects characterised by total deficiency of alveolar bone over the entire root length, have been reported to have lower success rate ranging from 27-37% (1-2). It is proposed that formation of long junctional epithelium during healing phase over the dehisced root surface may contribute to relatively lower success rate of such lesions (1, 3-4).

Successful treatment may, thus, depend not only on elimination of bacteria from the root canal system but also on preventing epithelial proliferation along denuded root surface. GTRtechniques with barrier membranes have been proposed as important adjunct in the management of endodontic-periodontal lesions. Such a membrane, when placed over a bony defect, may prevent the downgrowth of epithelial cells and provide an opportunity for the cells of the periodontal ligament and endosteum to regenerate the lost tissue (5-6).

Literature is replete with case reports and clinical studies (7-18) which demonstrate high success with GTR membrane, and advocate its use in apicomarginal defects (19-20). However, caution must be exercised in drawing any clinically relevant conclusions as none of these clinical studies had a control group. To the best of the investigator knowledge, only three experimental studies (21-23) have evaluated the utility of guided tissue regeneration in apicomarginal defects. While two of these have advocated use of the membrane in such lesions, one could not find any significant benefit of GTR.

Kim et al (24), in a recent prospective clinical study, reported 73.7% healing success by using calcium sulphate and collatape (resorbable collagen membrane) in periapical lesion with complete denudement of buccal bone plate (type F) and 63.6% success even if no membrane is used in E type of lesions. Recently, Song et al (25) also reported 70.4% healing success in apicomarginal defects without use of any GTR technique.These data suggest that there is possibility of healing of apicomarginal defects without use of any GTR technique, by using modern microsurgical techniques.

There is still inadequate information available regarding the suitability of GTR therapy in periradicular surgery in cases with apicomarginal defects. Only two randomized-clinical trials (17-18) have evaluated the healing response of GTR materials in treatment of apicomarginal defects. However, as in case of previously mentioned clinical studies, these too have not included any control group. Therefore, the purpose of this prospective, controlled clinical trial was to evaluate the role of collagen membrane as GTR material in healing of apicomarginal defects.

Materials and Methods

Subject Enrollment and Inclusion/Exclusion Criteria This clinical trial was conducted after obtaining ethical approval from the Institutional Ethics Board of Pandit Bhagwat Dayal Sharma University of Health Sciences, Rohtak. Forty study subjects were recruited from the pool of patients referred to the Department of Conservative Dentistry at Post Graduate Institute of Dental Sciences, Rohtak, India, between January 2012 and January 2013. The age of the patients ranged from 16 to 47 years. Eligibility criteria included apicomarginal communication confined to buccal aspect with a pocket depth (PD) of >6 mm and recurrent episodes of purulent discharge, teeth with negative response to vitality tests, with radiographic evidence of periapical radiolucencies, failed previous root canal treatment or retreatment at least 1 year previously, and adequate final restoration with no clinical evidence of coronal leakage. Teeth with vertical root fracture, resorptive processes extending to more than the apical third of the root, and subjects with chronic generalized periodontitis, systemic disease contraindicating surgical procedures, and conditions affecting rate of healing like diabetes and smoking were excluded from the study. All patients were duly informed of the nature of the study, the procedures involved and associated risks and benefits before obtaining their written consent. The minimum sample size was determined to be 15 patients in each treatment group on the basis of an error of α=0.05 and power at 0.80.

Preoperative Procedures and Primary Outcome Measurements After obtaining consent, the patients were thoroughly examined and clinical signs and symptoms were recorded carefully. Each patient received full mouth scaling and root planing, and, if needed, occlusal adjustments were carried out. The patients were then recalled after one week for baseline examination. All clinical periodontal measurements were performed by a same investigator (R.R). The clinical parameters recorded included periodontal PD, CAL and GMP. Each of these were measured on the buccal aspect of mesial and distal interproximal space and the mid buccal aspect of involved teeth (rounded off to the nearest mm) using a Williams O probe. Only the site with the deepest measurement at baseline was taken into consideration. PD was measured from the gingival margin to the base of the defect. The cemento-enamel junction (CEJ) or the apical border of the restoration, if the CEJ was not visible, was used as a reference for CAL & GMP measurement. The digital radiographs were taken with Kodak RVG 6000 (Kodak Digital Radiography System, Pt. Husada intra Care, Indonesia) using the Rinn (XCP Instruments, Elgin, IL) parallel device at 0, 3, 6, 9, and 12 months interval. Using CDR DICOM software (Schick CDR Technologies, Long Island City, NY), the digital x-ray images were divided into grid blocks, each with size of 1 mm2. Finally, the size of the lesion was calculated by counting the number of blocks with more than 50% area lying in the radiolucent lesion. Subjects were randomly assigned to the GTR membrane group or control group without stratification to eliminate any bias. Using an equal proportion allocation technique, sealed envelopes with assigned code were created by another investigator (S.T), which were then utilized for randomization of the subjects in the two given groups. It was further ensured that neither the surgeon, nor the patients were aware of the group allocation till the time of placement of membrane.

Surgical Techniques

All surgical procedures except for incision, flap elevation, and suturing, were performed under operating microscope (OPMI PICO; carl Zeiss, Gottingen, Germany) by the same operator (R.R). All the clinical procedures were performed using a standard surgical protocol reported in a previous study (18).

Briefly, a full-thickness mucoperiosteal flap was raised after deep anesthesia and osteotomy was performed. After debridement of the pathologic tissue, involved root was resected approximately 3 mm from the apex with a no. 170 tapered fissure bur under copious saline irrigation and hemostasis was achieved using cotton pellets soaked in 0.1% epinephrine (Jackson Lab (P) Ltd, Punjab, India). Then, the entire area of dehiscence along with the resected root surfaces was stained with the methylene blue and inspected with micromirrors (Hu-Friedy, Chicago, IL) under a high magnification of 26X to identify isthmuses, fins and other anatomic details of consequence. Root-end preparation with an approximate depth of 3 mm was made with S12-7D ultrasonic retrotips (Satelec) using a piezoelectric ultrasonic unit (P5 Booster,Suprasson Neutron; ActeonInc, Mt. Laurel, NJ). After ensuring the cleanness of the preparation, root-end filling was done with mineral trioxide aggregate (Pro Root; Retroplast Trading, Rorvig, Denmark).

In the GTR group, a bioresorbable collagen membrane (Healiguide, Advanced Biotech Products (P) Ltd., Encoll Corp., Fremont, CA, USA) was placed over the apicomarginal defect, covering 2-3mm of the healthy bone around all the margins. No membrane was placed in control group. Flap was carefully repositioned and then sutured with nonabsorbable 4-0 monofilament sutures. Traditional wound compression was avoided in GTR membrane group to prevent collapse of the membrane. Postoperatively, the patient was instructed to rinse his mouth twice daily with 0.2% chlorhexidine gluconate (Hexidine; ICPA health products ltd, India) for plaque control up to 10 days after surgery. The patient was recalled after 4 to 7 days for removal of sutures at the time of which the healing of the surgical site was checked and recorded.

Outcome Assessment

The radiographic examination was carried out every 3 months up to the period of 12 months using the same exposure parameters as baseline. Clinical evaluation was also done at the said intervals to look for any signs of failure. However, PD, CAL, and GMP were not measured until 12 months. Follow up radiographs were compared with baseline independently by two examiners (P.S, S.M) blinded to the group to which they belonged. Radiographic periapical healing was designated as complete, incomplete, uncertain, or unsatisfactory according to the criteria used by Rud et al (26) and Molven et al (27). The category was confirmed for data entry only when two examiners agreed on the same healing category. In case of discrepancy, the examiners sat together and discussed to arrive at a consensus. For statistical reasons, the results obtained were further dichotomized into success or failed cases. The criteria for success included the absence of clinical signs and symptoms, and complete or incomplete radiographic healing. Criteria for failed cases included those with any clinical signs or symptoms and/or radiographic evidence of uncertain or unsatisfactory healing.

Statistical Analysis

Data were presented as the mean ± standard deviation. Statistical tests performed were two tailed and interpreted at the 5% significance level. The statistical analyses of the ordinal data were carried out by using nonparametric methods. Mann-Whitney and Wilcoxon signed rank tests were used for unpaired and paired data, respectively. Chi-square test was utilized to evaluate dichotomous data. The interobserver reliability was analyzed with the Cohen kappa analysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria included apicomarginal communication confined to buccal aspect with a pocket depth (PD) of >6 mm and recurrent episodes of purulent discharge, teeth with negative response to vitality tests, with radiographic evidence of periapical radiolucencies, failed previous root canal treatment or retreatment at least 1 year previously, and adequate final restoration with no clinical evidence of coronal leakage

Exclusion Criteria:

* Teeth with vertical root fracture, resorptive processes extending to more than the apical third of the root, and subjects with chronic generalized periodontitis, systemic disease contraindicating surgical procedures, and conditions affecting rate of healing like diabetes and smoking were excluded from the study.

Ages: 16 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pocket depth | baseline to one year
Clinical attachment level | baseline to one year
Gingival margin position | baseline to one year
size of apical radiolucency | baseline to one year

SECONDARY OUTCOMES:
pain swelling sinus tract | base line to one year